CLINICAL TRIAL: NCT01795131
Title: Role of Vitamin B12 Supplementation During Pregnancy and Postpartum to Reduce Nutritional Anemia and Improve Immunity in Bangladeshi Women and Their Infants
Brief Title: Vitamin B12 Supplementation During Pregnancy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PR-09033
Record Dates: First submitted 2013-02-09; First posted 2013-02-20 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2009-07

CONDITIONS: Nutritional Anemia in Mothers.; Nutritional Anemia in Infants.
Keywords: Nutritional anemia; Vitamin B12; flu vaccine; immunity
MeSH Terms: conditions — Influenza, Human | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin B12 (Active Comparator): Supplementation group (N=60) that will receive 250 µg of vitamin B12 in addition to 60 mg of Fe and 400µg of folate.
  Interventions: Dietary Supplement: Vitamin B12
- Placebo (Placebo Comparator): Placebo group (N=60) that will receive placebo tablets and 60 mg of Fe and 400µg of folate daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B12
  Arms: Vitamin B12
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Nutritional anemia is a major public health problem among children and women in developing countries. Despite ongoing national program of supplementing pregnant women with iron-folate, prevalence of anemia is 39% among pregnant women and 78% among infants in Bangladesh. Vitamin B12 deficiency is a more prevalent cause of megaloblastic anemia than folate in many developing countries. This data raises the interest to address the role of vitamin B12 deficiency in nutritional anemia. Low dietary intake of animal products, a predominant source of vitamin B12 may cause anemia. Besides maintaining normal erythropoiesis, B12 is essential for immune function. However, no studies have evaluated the effect of maternal B12 supplementation on reduction of anemia and improving immunity of their infants. The investigators hypothesize that vitamin B12 supplementation plus iron-folate during pregnancy and 3-mo postpartum would: (a) Decrease anemia among mothers and infants; (b) Improve vaccine specific cellular and humoral immune responses among mothers; (c) Improve vaccine specific immunity in infants by passive transfer; (d) Improve DNA methylation and one-carbon metabolism in mother-child pairs; (e) Reduce antenatal/postnatal depression. Results from this study will guide and provide support to the policy makers to identify effective strategies to reduce nutritional anemia in population at risk.

The investigators aim to conduct a double-masked placebo controlled trial to investigate the added effect of vitamin B12 on the iron-folate supplementation among pregnant women. Anemic (Hb level <11.0 g/dl) mothers at 11-14 weeks of gestation will be randomized into two groups: supplement group will receive 250 ug vitamin B12 plus 400 ug folate and 60 mg iron; placebo group will receive folate and iron only. This daily supplementation will continue up to 3-mo postpartum. At 26-28 wk of gestation mothers will be given inactivated influenza vaccine. Data on anthropometric indices of mothers and children, birth size, infant growth and morbidity (mothers and children) throughout the study period will be recorded. 24-h dietary recall data will be collected from the mothers bimonthly throughout the study. Biochemical indicators of anemia including Hb, vitamin B12, ferritin, folate and α-glycoprotein (AGP) will be assessed in plasma of mothers (pre- and post-supplementation) and infants (cord blood and 3-months). Additional measurements include serum transferrin receptor (sTfR) in plasma and methyl malonic acid (MMA) and total homocysteine (tHcy) in the urine of mothers. Plasma vaccine specific antibody responses will be measured in mothers (pre- and post supplementation) and in infants (cord blood and 3-months). In breast milk, B12, folate and s-IgA will be determined. Genetic polymorphism (one-carbon metabolism) and DNA methylation will be studied in mothers and in cord blood.

DETAILED DESCRIPTION:
Study Area: A maternity clinic in Mirpur with substantial numbers of pregnant women enrolling each month (about 300-400/month) will be selected for recruitment of local pregnant women. The community in Mirpur has a low out-migration rate. Pregnant women attending the clinic at 11-14 weeks of gestation and planning to deliver at the clinic to ensure safe delivery will be selected. The structured service and standard antenatal care of the clinic for safe delivery and antenatal care will be provided to each study participant.

Study Population: Pregnant women (n=120) will be screened during 11-14 weeks of gestation. Infants (n=120) at 3 months of age.

Inclusion Criteria:

* Hb level in the range of 7.0-11 g/dL
* Age: 22-35 years
* Mothers at the beginning of second trimester (i.e. at 11-14 weeks of gestation)
* Willing to stay in Dhaka during pregnancy and willing to get admitted in the clinic for delivery
* Self-reported Last Menstrual Period (LMP) and urine pregnancy test will be used to determine the gestational age.

Exclusion Criteria:

* Women with severe anemia; hemoglobin concentration <7.0 g/dL
* History or presence of systemic disease
* H/O of previous complicated pregnancies or of pre-term delivery, abortion
* Receipt of influenza vaccine Definition: According to WHO, anemia is defined as a hemoglobin concentration <12 g/dL in adult women. Anemia is further categorized as mild (10-11.9 g/dL), moderate (7.0-9.9 g/dL) and severe (<7.0 g/dL).

Study design: A double-blind controlled trial; After informed consent is obtained, pregnant women will be randomly assigned either to Placebo group (N=60) that will receive 60 mg of Fe and 400µg of folate daily or Supplementation group (N=60) that will receive 250 µg of vitamin B12 in addition to 60 mg of Fe and 400µg of folate. A third party (GlaxoSmithKline, Bangladesh) will prepare and supply vitamin B12 or placebo capsule in bottles. The two capsules will be similar in appearance and taste. They will label the bottles as A and B. The responsible personnel from the Company will keep it confidential until the end of study. The capsule either A or B to be received by the 1st participant will be determined by a lottery, and thereafter every alternate participant will receive that capsule. The IDs of the participants will be given sequentially. The daily supplementation of iron-folate as well as of B12 will continue up to 3-months postpartum. At 26-28 weeks of gestation, all mothers will receive a single inactivated, trivalent influenza virus vaccine intramuscularly (IM). Standard inactivated trivalent influenza as recommended by WHO for the Northern Hemisphere will be obtained from commercial sources for this project (GlaxoSmithKline; Dresden, Germany). Field workers (FW) will deliver two weeks' dose of either placebo or supplements to mothers in person and will check the compliance by card and left over pills. The pregnant women will be clearly instructed about the times for their subsequent follow-up visits, and when followed up in respective homes they will be reminded of the dates.

Routine Service: The routine care provided by the clinic includes Hb measurement, physical examination (weight, blood pressure, pulse rate, abdominal check-up, fetal heart rate, ultrasonographic examination as necessary), counseling on diet, descriptions of normal procedures during pregnancy, associated potential complications, how and when to go to the clinic during such events etc. This service is provided by the clinic physician with assistance from the nurses.

Specimens: Fasting peripheral blood will be collected from mothers at 11 to 14 weeks of gestation, cord blood at delivery, colostrums within 24 hours and breast milk and peripheral blood from mothers after three months postpartum. Peripheral blood from infants will be collected at three months of age. Blood will be collected in anticoagulant (EDTA) coated tubes and layered on Ficoll-paque for density gradient centrifugation; plasma will be separated from the top and stored at -70ºC for later analysis. Peripheral blood mononuclear cells (PBMC) will be separated for studying cellular immune responses. Urine will be collected from mothers at 11 - 14 weeks of gestation and at three months. For gene based studies, the DNA samples will be delinked and the identity will be made anonymous according to the standard procedures.

Methods: Total hemoglobin (Hb) in whole blood will be measured by spectrophotometry using Drabakins Reagent (Sigma Diagnostics). Standardized blood smear stain will be used for evaluating megaloblastic anemia (presence of macroovalocytes and hypersegmented neutrophils). Ferritin, serum transferrin receptor (sTfR) and α-glycoprotein (AGP) will be measured in plasma by enzyme immune assays. Vitamin B12 and folate in plasma and vitamin B12 in breast milk will be assayed in Roche autoanalyzer Cobas e411. Urinary methyl malonic acid (MMA) will be measured by fluorescence detector assisted HPLC method (Sigma Diagnostics, St. Louis, MO. Briefly MMA will be extracted from urine sample with ethyl acetate. The extract is dried and derivatized with monodansylcadaverine and dicyclohexyl-carbodiimide prior to injection on the HPLC. Ethylmalonic acid will be used as an internal standard. Influenza vaccine-specific antibody responses (IgA, IgG) in plasma and colostrum/ breast milk [secretory IgA (s-IgA)] will be measured by ELISA. PBMC will be stimulated with Flu vaccine for blastogensis response. Genomic DNA methylation will be measured by the methyl acceptance assay based on the ability of isolated DNA to "accept" radiolabeled methyl groups from S-[3H-methyl] adenosylmethionine, using the bacterial CpG methyltransferase SssI. Total homocysteine (tHcy) will be measured in urine samples by using HPLC with fluorimetric detection in which Thiols in the column effluent are detected by a single gold-mercury electrode. NaBH4 is used as a reductant, and no derivatization of sample is required. Mutations in the ALPL, MTHFR C677T and FUT2 genes will be determined by PCR- RFLP assay and DNA sequencing. All these assays will be performed in the Nutritional Biochemistry Lab which has the facilities to determine the biochemical markers of anemia, vaccine specific antibody responses, DNA methylation and polymorphism assays.

Assessment of anthropometry and morbidity: Maternal anthropometrical measurements will be taken at the beginning of supplementation and monthly during the post supplementation period by trained FWs. Birth weight and recumbent length will be taken within 72 hours after birth and monthly measurements will be taken by FW up to 3 mo of age. At each visit (fortnightly), Field Research Assistant (FRA) will collect data from mothers on morbidity of mothers and their infants (e.g. diarrhoea, respiratory infections, skin diseases, assessment of severity of disease episodes) of the previous 7 days using structured questionnaires. The FRAs will inform the women about the times of the first and subsequent follow-up visits, and ensure if they have understood clearly. In addition, study participants will be contacted over cell phones when available to remind them about the visit dates. When followed up in respective homes, they will be reminded of the next visit dates.

Depression score: Participants will be interviewed on their mental status using the Centre for Epidemiological Studies-Depression (CES-D) questionnaire. The questionnaire contains 20 items comprising six major aspects of depression: depressed mood, hopelessness, worthlessness, fatigue, appetite and sleep disturbances. It was translated to Bengali and piloted in earlier studies and involves how the women felt during the preceding 7 days. It has been previously used in rural and urban Bangladeshi women (Hamadani, unpublished data) and found to correlate sensibly to children's growth and development. The FRAs will be extensively trained to interview the women and inter-observer reliabilities will be obtained before and during the study. The interview will be conducted twice at the homes of the women during FRAs' visits, first at baseline and at 3 mo postpartum. The data will be analyzed and interpreted by one of the co-investigators (JDH) who has knowledge and experience in dealing with this type of information.

Food security and dietary diversity: The effect of food insecurity on food intake, health and nutritional status has been observed in many developing countries showing significantly lower total daily per capita food expenditures in food-insecure households than food-secure households. Food insecurity was associated with maternal anxiety and depression, which can have strong negative influence on infant care practices including breastfeeding duration as well as child nutritional status. About half of the Bangladeshi population is food-insecure. Hunger and childhood malnutrition in Bangladesh are among the highest in the world. About 31% of the rural population in Bangladesh suffers from "chronic poverty" and about 19% of rural households cannot have "full three meals" a day. Thus, household food insecurity in relation to its enormous impact on health and nutritional status on human is a growing concern in Bangladesh. Household food security status and dietary diversity of the study participants (including maternal dietary energy, protein, vitamin B-12 and folate intake) will be assessed first, at the baseline when the pregnant women will be enrolled in the study and thereafter fortnightly throughout the study. USDA food composition database will be used for assessing vitamin B-12 intake. Any seasonal variation of the food security status will be assessed that might have significant impact on the outcome measures. Structured questionnaire on food security module will be used to measure household food security status. The FRAs will be trained to interview the women; they will take interviews when they make visits during the antenatal and postnatal periods at the home. The data will be analyzed and interpreted by one of the co-investigators (KKS) who has knowledge and experience in dealing with this type of information.

ELIGIBILITY:
Inclusion Criteria:

1. Hb level in the range of 7.0-11 g/dL
2. Age: 22-35 years
3. Mothers at the beginning of second trimester (i.e. at 11-14 weeks of gestation)
4. Willing to stay in Dhaka during pregnancy and willing to get admitted in the clinic for delivery
5. Self-reported Last Menstrual Period (LMP) and urine pregnancy test will be used to determine the gestational age.

Exclusion Criteria:

1. Women with severe anemia; hemoglobin concentration <7.0 g/dL
2. History or presence of systemic disease
3. H/O of previous complicated pregnancies or of pre-term delivery, abortion
4. Receipt of influenza vaccine

Ages: 22 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
a) Percent reduction in nutritional anemia among mothers (based on measurement of Hb, ferritin, sTfR, folate, B12 levels in plasma; urinary MMA and tHcy; B12 levels in breast milk.) | 24 months
  The investigators will determine the percentage of nutritional anemia in mothers by measuring Hb, ferritin, sTfR, B12 levels in plasma. They will also measure urinary MMA and tHcy and B12 levels in breast milk.
Increase in influenza vaccine specific cellular and humoral responses among mothers (blastogenesis and T cell phenotyping,serum IgA, and IgG). | 24 monnths
  Influenza vaccine-specific antibody responses (IgA, IgG) in plasma and colostrum/ breast milk [secretory IgA (s-IgA)] will be measured by ELISA. PBMC will be stimulated with Flu vaccine for blastogensis response.
Increase in influenza vaccine specific immunity in infants by passive transfer (vaccine specific IgG in cord blood and breast milk and IgA in children at 3 mo). | 24 months
  Influenza vaccine-specific antibody responses (IgA, IgG) in plasma and colostrum/ breast milk [secretory IgA (s-IgA)] will be measured by ELISA. PBMC will be stimulated with Flu vaccine for blastogensis response.
Percent reduction in nutritional anemia in infants (based on measurement of Hb, ferritin, B12 levels in plasma; | 24 months
  The investigators will determine the percentage of nutritional anemia in mothers by measuring Hb, ferritin, B12 levels in plasma.

SECONDARY OUTCOMES:
Effect of B12 status on DNA methylation and one-carbon metabolism in mother-child pairs. | 24 months
  Genomic DNA methylation will be measured by the methyl acceptance assay . Total homocysteine (tHcy) will be measured in urine samples by using HPLC with fluorimetric detection. Mutations in the ALPL, MTHFR C677T and FUT2 genes will be determined by PCR- RFLP assay and DNA sequencing.
Reduce depression scores | 24 months
  Participants will be interviewed on their mental status using the Centre for Epidemiological Studies-Depression questionnaire. The questionnaire contains 20 items comprising six major aspects of depression: depressed mood, hopelessness, worthlessness, fatigue, appetite and sleep disturbances. It has been previously used in rural and urban Bangladeshi women (J Hamadani) and found to correlate sensibly to children's growth and development. The interview will be conducted twice at the homes of the women first at baseline and at 3 mo postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Rubhana Raqib, Ph D, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Maternal and Child Health Training Institute, Dhaka, Bangladesh

REFERENCES:
- [Derived] Siddiqua TJ, Akhtar E, Haq MA, Shahab-Ferdows S, Hampel D, Islam S, Ahmed T, Allen LH, Raqib R. Effects of vitamin B12 supplementation on oxidative stress markers and pro-inflammatory cytokines during pregnancy and postpartum among Bangladeshi mother-child pairs. BMC Nutr. 2024 Jan 3;10(1):3. doi: 10.1186/s40795-023-00785-y. PMID 38172996